CLINICAL TRIAL: NCT04875468
Title: Clinical Outcomes of Bonded Monolithic Translucent Zirconia Crowns Using Two Different Compositions of Self-adhesive Resin Cements (Randomized Clinical Trial)
Brief Title: Clinical Outcomes of Bonded Monolithic Translucent Zirconia Crowns Using Two Different Compositions of Self-adhesive Resin Cements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diana Mostafa Habeb (Other)
Responsible Party: Sponsor-Investigator, Diana Mostafa Habeb, Assistant Lecturer of Fixed Prosthodontics, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28611222102086
Record Dates: First submitted 2021-04-30; First posted 2021-05-06 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Destructed Teeth Restored by Zirconia Crowns; Zirconia Crowns; Decayed, Missing, and Filled Teeth; Tooth Discoloration
Keywords: Marginal adaptation, patient satisfaction
MeSH Terms: conditions — Dental Caries; Tooth Discoloration; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zirconia crown cemented by adhesive resin cement (Active Comparator): MultiRein link adhesive resin cement (non MDP, non-calcium and fluoride releasing cement)
  Interventions: Other: Multilink adhesive resin cement
- Zirconia crown cemented by self-adhesive resin cement (Experimental): TheraCem self-adhesive resin cement (MDP, calcium and fluoride releasing cement)
  Interventions: Other: TheraCem self-adhesive resin cement

INTERVENTIONS:
Other: TheraCem self-adhesive resin cement — MDP, calcium and fluoride releasing cement for dental zirconia crowns
  Arms: Zirconia crown cemented by self-adhesive resin cement
Other: Multilink adhesive resin cement — (non MDP, non-calcium and fluoride releasing cement)
  Arms: Zirconia crown cemented by adhesive resin cement

SUMMARY:
The aim of the present study is to evaluate the clinical outcomes (marginal discoloration, marginal adaptation, gingival health, debonding and patient satisfaction) of translucent zirconia crowns bonded by TheraCem (MDP, calcium and fluoride releasing) self-adhesive resin cement compared to multilink self-adhesive resin cement.

DETAILED DESCRIPTION:
Clinical outcomes of bonded monolithic translucent zirconia crowns using two different compositions of self-adhesive resin cements (Randomized Clinical Trial)

Research question:

Will TheraCem self-adhesive resin cement (MDP, calcium and fluoride releasing cement) give better outcomes when bonding monolithic translucent zirconia crowns to tooth structure compared to Multilink self-adhesive resin cement (non MDP, non-calcium and fluoride releasing cement) in terms of marginal discoloration, marginal adaptation, gingival health, debonding and patient satisfaction?

PICOS:

P: Population: Patients requiring single zirconia crowns I: Intervention: TheraCem self-adhesive resin cement (MDP, calcium and fluoride releasing cement) C: Comparison: Multilink adhesive resin cement (non MDP, non-calcium and fluoride releasing cement)

O: Outcomes:

Outcomes Primary outcome Marginal discoloration using USPHS for 9 months Secondary outcomes 1. Marginal adaptation

2. patient satisfaction

Statement of the problem:

Bonding of zirconia restorations to tooth structures is still challenging. The success of the restoration may be affected by the type of cement used as it may affect marginal discoloration, marginal adaptation, gingival health, debonding and patient satisfaction. The effect of newly introduced TheraCem self-adhesive resin cement (MDP, calcium and fluoride releasing cement) on the clinical behavior of bonded translucent monolithic zirconia is not yet fully reported.

Aim of the study:

- The aim of the present study is to evaluate the clinical outcomes (marginal discoloration, marginal adaptation and patient satisfaction) of translucent zirconia crowns bonded by TheraCem (MDP, calcium and fluoride releasing) self-adhesive resin cement compared to multilink self-adhesive resin cement.

Research null hypothesis:

-There will be no difference in color stability, marginal adaptation and patient satisfaction of translucent zirconia crowns bonded either with TheraCem or Multilink self-adhesive resin cements.

Primary objective:

The Primary outcome: Marginal discoloration using USPHS Secondary outcomes: 1. Marginal adaptation 2. Patient satisfaction

Trial design:

Parallel group, two arms, with 1:1 ratio

Methods:

A) Participants, interventions, and outcomes

Study setting: This study will be carried out on patients enrolled from the Outpatient clinic in fixed prosthodontics clinic, Faculty of Dentistry, Cairo University.

Eligibility criteria:

Inclusion criteria:

All subjects are required to be:

1. From 18-50 years old, be able to read and sign the informed consent document.
2. Have no active periodontal or pulpal diseases, have teeth with good restorations
3. Psychologically and physically able to withstand conventional dental procedures
4. Patients with teeth problems indicated for single crowns:

   1. Badly decayed teeth
   2. Teeth restored with large filling restorations
   3. Endodontically treated teeth
   4. Malformed teeth
   5. Malposed teeth (Tilted, over-erupted, rotated, etc.)
   6. Spacing between teeth
5. Able to return for follow-up examinations and evaluation.

Exclusion criteria:

1. Patient less than 18 or more than 50 years
2. Patient with active resistant periodontal disease
3. Patients with poor oral hygiene and uncooperative patients
4. Pregnant women
5. Patients in the growth stage with partially erupted teeth
6. Psychiatric problems or unrealistic expectations

Interventions:

TheraCem (MDP containing - calcium and fluoride releasing self-adhesive resin cement).

Outcomes The outcomes will be assessed at the following time points

T0 = immediately after restoration delivery

Primary Marginal Discoloration Alpha (A): no discoloration (There is no visual evidence of marginal discoloration different from the color of the restorative material and from the color of the adjacement.

(visual inspection)

Bravo (B): discoloration without axial penetration (There is visual evidence of marginal discoloration at the junction of the tooth structure and the restoration, but the discoloration has not penetrated along the restoration in a pulpal direction.

(visual inspection)

Charlie (C): discoloration with axial penetration (There is visual evidence of marginal discoloration at the junction of the tooth structure and the restoration that has penetrated along the restoration in a pulpal direction. (visual inspection Secondary 1.Marginal Adaptation Alpha (A) No visible evidences of crevice along the margins; no catch or penetration of the explorer.

Bravo (B) Visible evidence of crevice and/or catch of explorer; no penetration of the explorer.

Charlie (C) Visible evidence of crevice and penetration of explorer 2.Patient satisfaction Numerical (discrete) ("0" unsatisfied - "10" satisfied)

Participant timeline:

- The patient will be treated in visits designated as follows:

Visit 1: Pre-operative records, face-to-face adherence reminder session, clinical, radiographic examination, intraoral photographs and primary impression (alginate impression*) for diagnostic cast construction.

Visit 2: Teeth preparation, secondary impression using addition silicone rubber base material† and temporary restoration‡.

Visit 3: Try in Visit 4: placement and permanent cementation of the final restoration.

* Marginal discoloration, color stability, marginal adaptation and patient satisfaction will be evaluated immediately after cementation.

Recall visits:

The same evaluators evaluated the participants during the recall appointments with a mirror and a sharp explorer at 3 months, 6 months, and 9 months. Periapical radiographs were made and postoperative data were collected and used as a documentation tool with the clinical photographs. Marginal adaptation, esthetics, patient satisfaction and clinical examination were assessed using USPH After delivering the crowns, the participants were asked to rate the level of the satisfaction with their restorations by using a 1 to 10 numeric rating scale (1=poor, 5=acceptable, 10=excellent) at 3 months, 6 months and 9 months. Mean, standard deviation and 95% confidence interval for the mean were used to summarize patient satisfaction.

Data collection methods:

Primary outcome: Marginal discoloration will be assessed by using HSPHS criteria Secondary outcomes: 1. Marginal adaptation will be assessed using the modified USPHS criteria.

2. Patient satisfaction will be assessed by using normal scores numerical score from 1 to 10 (1=poor, 5=acceptable, 10=excellent)

ELIGIBILITY:
Inclusion Criteria:

* All subjects are required to be:

  1. From 18-50 years old, be able to read and sign the informed consent document.
  2. Have no active periodontal or pulpal diseases, have teeth with good restorations
  3. Psychologically and physically able to withstand conventional dental procedures
  4. Patients with teeth problems indicated for single crowns:

     1. Badly decayed teeth
     2. Teeth restored with large filling restorations
     3. Endodontically treated teeth
     4. Malformed teeth
     5. Malposed teeth (Tilted, over-erupted, rotated, etc.)
     6. Spacing between teeth
  5. Able to return for follow-up examinations and evaluation.

Exclusion Criteria:

* 1. Patient less than 18 or more than 50 years 2. Patient with active resistant periodontal disease 3. Patients with poor oral hygiene and uncooperative patients 4. Pregnant women 5. Patients in the growth stage with partially erupted teeth 6. Psychiatric problems or unrealistic expectations

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Marginal discoloration | 9 months
  Alpha (A): no discoloration (There is no visual evidence of marginal discoloration different from the color of the restorative material and from the color of the adjacement.
  (visual inspection)
  Bravo (B): discoloration without axial penetration (There is visual evidence of marginal discoloration at the junction of the tooth structure and the restoration, but the discoloration has not penetrated along the restoration in a pulpal direction.
  (visual inspection)
  Charlie (C): discoloration with axial penetration (There is visual evidence of marginal discoloration at the junction of the tooth structure and the restoration that has penetrated along the restoration in a pulpal direction. (visual inspection

SECONDARY OUTCOMES:
Marginal Adaptation | 9 months
  Alpha (A) No visible evidences of crevice along the margins; no catch or penetration of the explorer.
  Bravo (B) Visible evidence of crevice and/or catch of explorer; no penetration of the explorer.
  Charlie (C) Visible evidence of crevice and penetration of explorer
Patient satisfaction | 9 months
  Numerical (discrete) ("0" unsatisfied - "10" satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Giza Governorate, Egypt